CLINICAL TRIAL: NCT04956393
Title: Proof-of-Concept of the SOAR (Stop OsteoARthritis) Program: A Randomized Delayed-Control Trial
Brief Title: The SOAR (Stop OsteoARthritis) Program Proof-of-Concept Study
Acronym: SOARPOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: The Arthritis Society, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Jackie Whittaker, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB# H21-01491
Record Dates: First submitted 2021-06-23; First posted 2021-07-09 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Arthritis; Osteoarthritis; Arthritis Knee; Osteo Arthritis Knee; Knee Injuries; Anterior Cruciate Ligament Tear; Meniscus Tear
Keywords: Randomized delayed control trial; Knee health; Knee injury; Sport injury; Knee muscle; Self-efficacy; Quality of life; Osteoarthritis
MeSH Terms: conditions — Arthritis; Osteoarthritis; Knee Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate SOAR Program (Experimental): Participants with a past sport-related knee injury randomized to the 'immediate intervention' group will complete an 8-week (weeks 1-8) SOAR program (Knee Camp, home-based exercise-therapy and physical activity with tracking, weekly 1:1 physiotherapist counseling sessions, and optional weekly group-based exercise classes) followed by an additional 8 weeks (weeks 10-17) of home-based exercise-therapy and physical activity with tracking, weekly 1:1 PT counseling sessions, and optional weekly group-based exercise classes. Consented trained physiotherapists will deliver the SOAR program throughout the study period to one or more immediate SOAR group knee injury participants.
  Interventions: Behavioral: Immediate 8-Week SOAR Program
- Delayed SOAR Program (Other): Participants with a past sport-related knee injury randomized to the 'delayed intervention' group will have a 9-week unstandardized delay before completing an 8-week SOAR program (weeks 10-17). During the delay (weeks 1-9) the delay comparison intervention will be unstandardized to reflect usual care in Canada. After the 9-week delay, these participants will complete an 8-week (weeks 10-17) SOAR program (Knee Camp, home-based exercise-therapy and physical activity with tracking, weekly 1:1 PT counseling sessions, and an optional weekly group-based exercise classes). Consented trained physiotherapists will deliver the SOAR program from week 10 to week 17 to one or more delayed SOAR group knee injury participants.
  Interventions: Behavioral: Delayed 8-Week SOAR Program

INTERVENTIONS:
Behavioral: Immediate 8-Week SOAR Program — This is an 8-week, virtually delivered, exercise-based, knee health program delivered to knee injury participants by trained physiotherapists. The program has 3 components:
  1. Knee Camp: This includes an interactive education session about knee health, 1:1 knee exam, and 1:1 counseling session to identify Specific, Measurable, Attainable, Relevant, and Time-bound (SMART) weekly home-based exercise-therapy and physical activity goals, Participants are asked to wear Fitbit's® 24-hours/day.
  2. Weekly Home-based Exercise-Therapy and Physical Activity, with Tracking: At home, participants work to meet their exercise-therapy and physical activity goals. Exercises are tracked with an online bespoke form and activity, with a Fitbit.
  3. Weekly PT-guided Exercise-Therapy and Physical Activity Counseling Sessions: Each week participants will attend a 1:1 virtual physiotherapist counseling session to modify SMART goals and have the option to attend a group exercise class.
  Arms: Immediate SOAR Program
Behavioral: Delayed 8-Week SOAR Program — This is an 8-week, virtually delivered, exercise-based, knee health program delivered to knee injury participants by trained physiotherapists. The program has 3 components:
  1. Knee Camp: This includes an interactive education session about knee health, 1:1 knee exam, and 1:1 counseling session to identify Specific, Measurable, Attainable, Relevant, and Time-bound (SMART) weekly home-based exercise-therapy and physical activity goals, Participants are asked to wear Fitbit's® 24-hours/day.
  2. Weekly Home-based Exercise-Therapy and Physical Activity, with Tracking: At home, participants work to meet their exercise-therapy and physical activity goals. Exercises are tracked with an online bespoke form and activity, with a Fitbit.
  3. Weekly PT-guided Exercise-Therapy and Physical Activity Counseling Sessions: Each week participants will attend a 1:1 virtual physiotherapist counseling session to modify SMART goals and have the option to attend a group exercise class.
  Arms: Delayed SOAR Program

SUMMARY:
Adolescents and young adults who hurt their knees playing sports or doing recreational activities can develop joint damage, muscle weakness, inactivity, and weight gain which might lead to an increased risk of osteoarthritis (OA), a disabling joint condition in their later lives. Despite knowing that muscles and joints benefit from exercise, there is no proven exercise-based treatments to delay or even halt the onset of OA after a knee joint injury.

The current study will assess if a physiotherapist-guided intervention called Stop OsteoARthritis (SOAR) improves knee muscle strength, physical inactivity, knee-related self-efficacy, and knee-related quality of life in people at risk for osteoarthritis due to a past knee injury. A total of 70 former knee injury participants will be randomly assigned to two groups. One group will immediately start a 16-week SOAR program, while the second will wait for 9-weeks before starting an 8-week SOAR program. Trained physiotherapists will deliver the SOAR program with videoconferencing. The study hypothesis is that participating in the 8-Week SOAR program will improve the knee muscle strength, physical activity levels, knee-related self-efficacy and knee-related quality of life in people discharged from regular healthcare after a sports knee injury. The findings will help researchers understand the ideal length of the program for a future clinical trial in real-world settings.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to evaluate a novel, virtually delivered, PT-guided, knee health program (Stop OsteoARthritis - SOAR) for people who have been discharged from regular healthcare after a sports knee injury.

Objectives:

1. The primary objective of the study is to assess the efficacy of an 8-week SOAR program to improve knee muscle strength measured by computerized dynamometry (primary outcome and daily average moderate to vigorous physical activity measured by Tri-axial Accelerometer (secondary outcome), self-reported knee-specific self-efficacy (secondary outcome), and self-reported knee-related quality of life (secondary outcome) in people discharged from regular care after sports knee trauma. Several exploratory outcomes will also be assessed to inform the design of a future clinical trial.
2. A secondary objective of this study is to evaluate the feasibility of a protocol for a future full-scale clinical trial to assess the effectiveness and implementation of SOAR. Both SOAR program and study protocol implementation and practicality outcomes will be collected.
3. A third objective of this study is to inform the optimal length of the SOAR program.
4. A fourth, exploratory objective, of this study, is to explore the experiences of stakeholders (i.e., knee injury participants and physiotherapists) to inform future implementation.

Research Design:

This is a proof-of-concept, two-armed, open-label, randomized delayed control trial with embedded 1:1 interviews. In this design, randomization determines when the intervention is provided (immediate or 9-week delay). Consenting eligible knee injury participants will be randomly allocated in a 1:1 ratio to immediate intervention (experimental) or delayed intervention (control) groups using a computer-generated sequence of random numbers. Consenting eligible and physiotherapists will complete Brief Action Planning certification and SOAR training before delivering the SOAR program virtually to the knee injury participants.

The immediate study group will be complete an 8-week (weeks 1-8) SOAR program (Knee Camp, home-based exercise-therapy and physical activity with tracking, weekly 1:1 PT counseling sessions, and optional weekly group-based exercise classes) followed by an additional 8 weeks (weeks 10-17) of home-based exercise-therapy and physical activity with tracking, weekly 1:1 PT counseling sessions, and optional weekly group-based exercise classes. In contrast, after a 9-week delay, the delayed study group will complete an 8-week (weeks 10-17) intervention (Knee Camp, home-based exercise-therapy and physical activity with tracking, weekly 1:1 PT counseling sessions, and optional weekly group-based exercise classes).

Knee injury participant outcomes will be evaluated at baseline (T0), 9-weeks (T1-primary endpoint to assess efficacy), and 18-weeks (T2- endpoint to inform optimal intervention length).

Physiotherapist participants will be evaluated prior to training, immediately after training, and after they have delivered the SOAR program to all knee injury participants that they have been assigned in the study.

Statistical Analysis:

Descriptive statistics will be calculated for all demographic variables, and observed differences (sex, prior injury, injury type, prior treatment, etc.) considered when interpreting findings. Randomization integrity will be monitored. Outcomes will be disaggregated by sex and gender, and mean differences between T0 and T1, and T1 and T2 described by the study group. Intention-to-treat analyses will be conducted. Generalized linear mixed-effects regression models for longitudinal data (95%CI), controlling for the blocking effect, will estimate the effect of an 8-week intervention (IG T1-T0 versus DG T1-T0, and DG T2-T1 versus T1-T0) and the delay (IG T1-T0 versus DG T2-T1) for the primary outcome (Figure 2).

In addition, two exploratory analyses will be conducted. To inform the optimal intervention length for the future clinical trial, a longitudinal mixed-effects model will be used to examine the intervention effect at 16-week. This model will include the following fixed effects: 1) the randomization group indicator for baseline difference; 2) indicator variables for follow-up assessment time points (9-week and 18-week) to account for secular trend, and; 3) indicator variables for the lengths of time since intervention initiation (9-week or 18-week) to estimate effects after these time intervals. The model will also include participant-specific random effects to account for repeated measures. To inform the most meaningful muscle function outcome for the future clinical trial linear regression (95%CI) models, adjusted for age and sex, will be used to identify differences in the association between various aspects of knee extensor muscle function (torque, power, rate of force development), and composite self-reported knee symptoms and function score.

Interview recordings with knee injury participants and physiotherapist participants will be transcribed verbatim and de-identified. Using a constant comparative approach data will be coded and categories developed by comparing and determining meaningful patterns across codes. High-order themes will illuminate the relationship between categories. Uniqueness in experience by gender will be explored and if identified, data will be reanalyzed in gender sub-groups. A detailed audit of analytic decisions will be kept.

ELIGIBILITY:
Inclusion Criteria:

Knee Injury Participant Inclusion Criteria:

1. 16-35 years of age
2. Currently live in British Columbia, Canada
3. Experienced a sport-related intra-articular knee injury (i.e., clinical diagnosis of ligament, meniscal, or other intra-articular tibio- or patello-femoral trauma) that required both medical consultation (i.e., physician, physiotherapist, chiropractor, surgeon, or athletic therapist) and disrupted regular sports participation (missed at least one training session or competition) 12-36 months previously.18
4. Are currently not receiving ongoing health care related to the past knee injury and have no scheduled surgical procedures (any part of the body) that would interfere with exercise during the study.
5. Have daily access to an email address and a computer with internet
6. Are willing to wear an activity tracker during the study

Physiotherapist Participant Inclusion Criteria:

1. Registered physiotherapist
2. Able to communicate in English
3. Have an email address and daily access to a computer with internet service

Exclusion Criteria:

Knee Injury Participant Exclusion Criteria:

1. Inability to communicate in English
2. Previous physician diagnosis of index knee osteoarthritis
3. Inflammatory arthritis or systemic condition
4. Lower limb injury, surgery, or intra-articular injection in the past 6-months
5. Current pregnancy
6. Have a pacemaker or other internal medical device

Physiotherapist Participant Exclusion Criteria:

1. Do not hold a license to practice physiotherapy
2. Unable to communicate in English
3. Do not have an email address or daily access to a computer with internet service

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Change in Knee Extensor Strength over 9-weeks (knee injury participants) | Change from baseline knee extensor muscle strength at 9-weeks
  A computerized dynamometer (Biodex®) will be used to assess and calculate normalized peak concentric knee extension (quadriceps muscle) isokinetic torque (Nm/kg) at 90 degrees/seconds over 0-100 degrees of knee flexion. After a five-minute stationary cycling warm-up, participants will be seated with straps secured across their hips and chest. After three practice trials and a 30-second rest, participants will be instructed to straighten and bend their knee as hard as they can for three repetitions. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle strength.

SECONDARY OUTCOMES:
Change in Daily Average Moderate to Vigorous Physical Activity over 9-weeks (knee injury participants) | Change from baseline daily average moderate to vigorous physical activity at 9-weeks
  A small, lightweight hip worn wearable triaxial accelerometer (ActiGraph GT3X®) will be used to assess physical activity. Participants will be asked to wear this device (attached via an elastic belt around their waist), for a period of 7 consecutive days removing only for bathing/swimming activities. The average number of 10-minute moderate-to-vigorous physical activity bouts over the 7-day period will be calculated. Accelerometry is a valid measure of physical activity in youth and young adult populations.
Change in Self-reported Knee-specific Self-Efficacy over 9-weeks (knee injury participants) | Change from baseline knee-specific self-efficacy at 9-weeks
  A 19 item questionnaire (the Knee Self-efficacy Scale) will be used to measure self-reported knee-specific self-efficacy. Each item is scored on an 0-10-point Likert scale, with 0 indicating no knee-related self-efficacy and 10 indicating full knee-related self-efficacy. Individual item scores are summed and divided by 19 to produce a total score ranging from 0-10 (0 representing poor knee-related self-efficacy and 10 representing full knee-related self-efficacy). The total time for this questionnaire is 3 minutes. The Knee Self-efficacy Scale is a valid and reliable measure of knee-specific self-efficacy in individuals with a sport-related knee injury in the past five years.
Change in Self-reported Knee-related Quality of Life over 9-weeks (knee injury participants) | Change from baseline knee-related quality of life at 9-weeks
  A 5 item subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be used to measure self-reported knee-related quality of life. Each item is scored on an 0-10-point Likert scale, with 0 indicating no knee-related quality of life and 10 indicating full knee-related quality of life. Individual item scores are summed and transformed to a score out of 100 (0 representing poor knee-related quality of life and 100 representing full knee-related quality of life). The total time for this questionnaire is 3 minutes. The KOOS knee-related quality of life sub-scale is a valid and reliable patient-reported outcome measure across multiple patient populations, including at various timepoints after knee trauma

OTHER OUTCOMES:
Change in Knee Extensor Strength over 18-weeks (knee injury participants) | Change from baseline knee extensor muscle strength at 18-weeks
  A computerized dynamometer (Biodex®) will be used to assess and calculate normalized peak concentric knee extension (quadriceps muscle) isokinetic torque (Nm/kg) at 90 degrees/seconds over 0-100 degrees of knee flexion. After a five-minute stationary cycling warm-up, participants will be seated with straps secured across their hips and chest. After three practice trials and a 30-second rest, participants will be instructed to bend and straighten their knee as hard and as fast as they can for three repetitions. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle strength.
Change in Daily Average Moderate to Vigorous Physical Activity over 18-weeks (knee injury participants) | Change from baseline daily average moderate to vigorous physical activity at 18-weeks
  A small, lightweight hip worn wearable triaxial accelerometer (ActiGraph GT3X®) will be used to assess physical activity. Participants will be asked to wear this device (attached via an elastic belt around their waist), for a period of 7 consecutive days removing only for bathing/swimming activities. The average number of 10-minute moderate-to-vigorous physical activity bouts over the 7-day period will be calculated. Accelerometry is a valid measure of physical activity in youth and young adult populations.
Change in Self-reported Knee-specific Self-Efficacy over 18-weeks (knee injury participants) | Change from baseline knee-specific self-efficacy at 18-weeks
  A 19 item questionnaire (the Knee Self-efficacy Scale) will be used to measure self-reported knee-specific self-efficacy. Each item is scored on an 0-10-point Likert scale, with 0 indicating no knee-related self-efficacy and 10 indicating full knee-related self-efficacy. Individual item scores are summed and divided by 19 to produce a total score ranging from 0-10 (0 representing poor knee-related self-efficacy and 10 representing full knee-related self-efficacy). The total time for this questionnaire is 3 minutes. The Knee Self-efficacy Scale is a valid and reliable measure of knee-specific self-efficacy in individuals with a sport-related knee injury in the past five years.
Change in Self-reported Knee-related Quality of Life over 18-weeks (knee injury participants) | Change from baseline knee-related quality of life at 18-weeks
  A 5 item subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be used to measure self-reported knee-related quality of life. Each item is scored on an 0-10-point Likert scale, with 0 indicating no knee-related quality of life and 10 indicating full knee-related quality of life. Individual item scores are summed and transformed to a score out of 100 (0 representing poor knee-related quality of life and 100 representing full knee-related quality of life). The total time for this questionnaire is 3 minutes. The KOOS knee-related quality of life sub-scale is a valid and reliable patient-reported outcome measure across multiple patient populations, including at various timepoints after knee trauma
Change in Self-reported Knee-related Symptoms over 9-weeks (knee injury participants) | Change from baseline knee-related symptoms at 9-weeks
  The 8 and 18 item symptom and pain subscales of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be used to measure self-reported knee-related symptoms. Each item is scored on an 0-10-point Likert scale, with 0 indicating a high degree of symptoms and 10 indicating no symptoms. Individual item scores are summed and transformed to a score between 0 and 100, with higher scores indicating a better outcome (i.e., fewer knee-related symptoms). The total time for this questionnaire is 3 minutes. The KOOS knee-related symptoms sub-scale is a valid and reliable patient-reported outcome measure across multiple patient populations, including at various timepoints after knee trauma.
Change in Self-reported knee-related Sport and Recreation Function over 9-weeks (knee injury participants) | Change from baseline knee-related sport and recreation function at 9-weeks
  The 17 and 5 item function in daily living and function in sport and recreation subscales of the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire will be used to measure self-reported knee-related symptoms. Each item is scored on an 0-10-point Likert scale, with 0 indicating no knee-related sport and recreation function and 10 indicating full knee-related sport and recreation function. Individual item scores are summed and transformed to a score out of 100 (0 representing poor knee-related sport and recreation function and 100 representing full knee-related sport and recreation function). The total time for this questionnaire is 3 minutes. The KOOS knee-related sport and recreation function sub-scale is a valid and reliable patient-reported outcome measure across multiple patient populations, including at various timepoints after knee trauma.
Change in Self-reported Overall Function over 9-weeks (knee injury participants) | Change from baseline self-reported overall function at 9-weeks
  The 3 item Patient Specific Functional Scale will be used to identify, quantify and assess changes in functional limitations that are most relevant to participants. This scale prompts participants to identify three activities important to them and rate their ability to perform each activity on a 10-point numerical rating scale. Individual scale scores are summed and transformed to a 0-100 scale with higher scores indicating better outcomes. The total time for this questionnaire is 3 minutes. The Patient-Specific Functional Scale is valid and reliable for use in persons with a knee injury.
Change in Self-reported Physical Activity over 9-weeks (knee injury participants) | Change from baseline self-reported physical activity at 9-weeks
  The 4 item Godin Leisure Time Questionnaire will be used to measure self-reported physical activity. Using the number of 15-minute bouts of mild, moderate, and strenuous physical activity a participant engages in over a typical seven-day period weekly metabolic equivalents of physical activity are calculated. The total time for this questionnaire is 1 minute. The Godin Leisure Time Questionnaire has been validated to assess physical activity.
Change in Self-reported Perceived Self-care over 9-weeks (knee injury participants) | Change from baseline self-reported perceived self-care at 9-weeks
  The 12 item Partner in Health Scale will be used to measure perceived self-care (active involvement to self-manage a chronic condition). Each item is scored on a 0-9 point Likert scale. Scores on individual items are summed to produce a total score ranging between 0 and 96, with 0 representing no perceived self-management and 96 representing full perceived self-management. The total time for this questionnaire is 3 minutes. The Partner in Health Scale is valid and reliable across numerous chronic conditions.
Change in Self-reported Fear of Movement and Re-injury over 9-weeks (knee injury participants) | Change from baseline self-reported fear of movement and re-injury at 9-weeks
  The 11 item Tampa Scale of Kinesiophobia will be used to measure self-reported fear of movement and re-injury. Each item is scored on a 0-4 point Likert-scale, with 0 indicating no fear of movement and 4 indicating greater fear of movement. The item scores are summed to produce a total score ranging between 0 and 44, with higher values indicating a higher degree of fear of movement. The total time for this questionnaire is 3 minutes. The Tampa Scale of Kinesiophobia has evidence of known-group validity (scores discriminated between athletes who returned and did not return to pre-injury sports participation level after knee trauma).
Change in Self-reported Perceived Social Support from family and friends over 9-weeks (knee injury participants) | Change from baseline self-reported perceived social support from family and friends at 9-weeks
  The 12 item Multi-Dimensional Scale of Perceived Support will be used to measure perceived support from family, friends, and significant others. Each item is scored on a 0-7 point Likert scale, with 0 representing poor perceived support and 7 representing greater perceived support. Individual item scores are summed and divided by 12 to produce a total score ranging between 0 and 7 with higher scores indicating higher levels of perceived support. The total time for this questionnaire is 3 minutes. The Multi-Dimensional Scale of Perceived Support is reliable and valid across diverse general populations including adolescents.
Change in Self-reported Perceived Social Support from Sport and Recreation Community over 9-weeks (knee injury participants) | Change from baseline self-reported perceived social support from the sport and recreation community 9-weeks
  The 16 item Perceived Available Social Support Questionnaire will be used to assess perceived support from the sporting or recreational community. Each item is scored on a 0-4 point Likert scale, with 0 representing poor perceived support and 4 representing greater perceived support. Individual item scores are summed and divided by 16 to produce a total score ranging from 0 to 4, with higher scores indicating higher levels of perceived support. The total time for this questionnaire is 3 minutes. The Perceived Available Social Support Questionnaire is a valid and reliable measure of self-reported perceived support for sporting populations.
Change in Knee Flexor Strength over 9-weeks (knee injury participants) | Change from baseline knee flexor muscle strength at 9-weeks
  A computerized dynamometer (Biodex®) will be used to assess and calculate normalized peak concentric knee flexor (hamstring muscles) isokinetic torque (Nm/kg) at 90 degrees/seconds over 0-100 degrees of knee flexion. After a five-minute stationary cycling warm-up, participants will be seated with straps secured across their hips and chest. After three practice trials and a 30-second rest, participants will be instructed to straighten and bend their knee as hard as they can for three repetitions. The total time for this test is 10 minutes (assessed in conjunction with normalized peak knee extension torque). Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle strength.
Change in Knee Extension Power over 9-weeks (knee injury participants) | Change from baseline knee extensor muscle power at 9-weeks
  A computerized dynamometer (Biodex®) will be used to assess and calculate knee extension power (Watts). After completing the protocol for normalized peak concentric knee extension and flexion torque the participants' knee joint will be fixed in 60 degrees of sagittal plane flexion. After three practice trials and a 30-second rest, participants will be instructed to straighten their knee as hard and as fast as they can for five seconds. This will be repeated five times with a 30-second rest period between each repetition. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle power.
Change in Knee Flexion Power over 9-weeks (knee injury participants) | Change from baseline knee flexor muscle power at 9-weeks
  A computerized dynamometer (Biodex®) will be used to assess and calculate knee flexion power (Watts). After completing the protocol for normalized peak concentric knee extension and flexion torque the participants' knee joint will be fixed in 60 degrees of sagittal plane flexion. After three practice trials and a 30-second rest, participants will be instructed to bend their knee as hard and as fast as they can for five seconds. This will be repeated five times with a 30-second rest period between each repetition. The total time for this test is 10 minutes. Computerized dynamometry (Biodex®) is a reliable, valid, relevant, and recommended measure of muscle power.
Change in Hop function over 9-weeks (knee injury participants) | Change from baseline hop function at 9-weeks
  Single leg hop function will be measured using the 6-meter timed hop test. Participants are asked to hop forward with the goal of covering a 6-meter distance as quickly as they can. Two practice trials will be completed on each limb, starting with the unaffected side to familiarize participants with the task. Participants will then complete two test trials on each limb, starting again with the unaffected side. The time (seconds) required to hop the 6-m distance will be recorded. This protocol will take 10 minutes. The 6-m timed hop is clinically applicable and reliable.
Change in Fat Mass Index over 9-weeks (knee injury participants) | Change in fat mass index over 9-weeks (knee injury participants)
  Fat mass index (kg/m2) will be measured with Bioelectrical Impedance (Tanita Body Composition Analyzer, Model TBF-300A, Tanita Inc., USA). Participants will stand barefoot on the bioelectrical impedance platform during which the resistance to the flow of this single, high frequency alternating electrical current (500 A at 50 kHz) will be measured. Bioelectrical Impedance is a feasible method for assessing and tracking body composition in clinical settings and has been shown to be valid and reliable in child, youth, and adult populations. This test will take 5 minutes to complete. The device will be calibrated prior to each scan (according to the manufacturer's protocol).
Perspectives of the intervention at 18-weeks (knee injury participants) | Interviews will take place at 18-weeks
  At the end of the study, semi-structured 1:1 interviews will be conducted with a sub-sample of 15-20 knee injury participants. Using an inductive approach and interview guide, participants will be asked open-ended queries about their experiences with the intervention (SOAR program). Interviews will last approximately 45 minutes.
Change in confidence to deliver the intervention over 18-weeks (physiotherapist participants) | Change in confidence to deliver the intervention at 18-weeks
  A bespoke online survey will assess physiotherapists' overall confidence to deliver the intervention (SOAR program) including Brief Action Planning, SMART goal setting, and virtual physiotherapy delivery. Participants will be asked to rate their overall confidence on a 0-10 point numerical rating scale where 0 represents no confidence and 10 represents full confidence. The score will be transformed to a score between 0 and100, with higher scores indicating higher confidence. The survey will take 3 minutes to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Jackie L Whittaker, PhD, PT, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Safiri S, Kolahi AA, Smith E, Hill C, Bettampadi D, Mansournia MA, Hoy D, Ashrafi-Asgarabad A, Sepidarkish M, Almasi-Hashiani A, Collins G, Kaufman J, Qorbani M, Moradi-Lakeh M, Woolf AD, Guillemin F, March L, Cross M. Global, regional and national burden of osteoarthritis 1990-2017: a systematic analysis of the Global Burden of Disease Study 2017. Ann Rheum Dis. 2020 Jun;79(6):819-828. doi: 10.1136/annrheumdis-2019-216515. Epub 2020 May 12. PMID 32398285
- [Background] March LM, Bachmeier CJ. Economics of osteoarthritis: a global perspective. Baillieres Clin Rheumatol. 1997 Nov;11(4):817-34. doi: 10.1016/s0950-3579(97)80011-8. PMID 9429738
- [Background] Yu D, Jordan KP, Bedson J, Englund M, Blyth F, Turkiewicz A, Prieto-Alhambra D, Peat G. Population trends in the incidence and initial management of osteoarthritis: age-period-cohort analysis of the Clinical Practice Research Datalink, 1992-2013. Rheumatology (Oxford). 2017 Nov 1;56(11):1902-1917. doi: 10.1093/rheumatology/kex270. PMID 28977564
- [Background] Roos EM, Arden NK. Strategies for the prevention of knee osteoarthritis. Nat Rev Rheumatol. 2016 Feb;12(2):92-101. doi: 10.1038/nrrheum.2015.135. Epub 2015 Oct 6. PMID 26439406
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Snoeker B, Turkiewicz A, Magnusson K, Frobell R, Yu D, Peat G, Englund M. Risk of knee osteoarthritis after different types of knee injuries in young adults: a population-based cohort study. Br J Sports Med. 2020 Jun;54(12):725-730. doi: 10.1136/bjsports-2019-100959. Epub 2019 Dec 11. PMID 31826861
- [Background] Fernandes GS, Parekh SM, Moses J, Fuller C, Scammell B, Batt ME, Zhang W, Doherty M. Prevalence of knee pain, radiographic osteoarthritis and arthroplasty in retired professional footballers compared with men in the general population: a cross-sectional study. Br J Sports Med. 2018 May;52(10):678-683. doi: 10.1136/bjsports-2017-097503. Epub 2017 Nov 3. PMID 29101102
- [Background] Gianotti SM, Marshall SW, Hume PA, Bunt L. Incidence of anterior cruciate ligament injury and other knee ligament injuries: a national population-based study. J Sci Med Sport. 2009 Nov;12(6):622-7. doi: 10.1016/j.jsams.2008.07.005. Epub 2008 Oct 2. PMID 18835221
- [Background] Emery C, Tyreman H. Sport participation, sport injury, risk factors and sport safety practices in Calgary and area junior high schools. Paediatr Child Health. 2009 Sep;14(7):439-44. doi: 10.1093/pch/14.7.439. PMID 20808471
- [Background] Watt FE, Corp N, Kingsbury SR, Frobell R, Englund M, Felson DT, Levesque M, Majumdar S, Wilson C, Beard DJ, Lohmander LS, Kraus VB, Roemer F, Conaghan PG, Mason DJ; Arthritis Research UK Osteoarthritis and Crystal Disease Clinical Study Group Expert Working Group. Towards prevention of post-traumatic osteoarthritis: report from an international expert working group on considerations for the design and conduct of interventional studies following acute knee injury. Osteoarthritis Cartilage. 2019 Jan;27(1):23-33. doi: 10.1016/j.joca.2018.08.001. Epub 2018 Aug 18. PMID 30125638
- [Background] Toomey CM, Whittaker JL, Nettel-Aguirre A, Reimer RA, Woodhouse LJ, Ghali B, Doyle-Baker PK, Emery CA. Higher Fat Mass Is Associated With a History of Knee Injury in Youth Sport. J Orthop Sports Phys Ther. 2017 Feb;47(2):80-87. doi: 10.2519/jospt.2017.7101. PMID 28142363
- [Background] Whittaker JL, Toomey CM, Nettel-Aguirre A, Jaremko JL, Doyle-Baker PK, Woodhouse LJ, Emery CA. Health-related Outcomes after a Youth Sport-related Knee Injury. Med Sci Sports Exerc. 2019 Feb;51(2):255-263. doi: 10.1249/MSS.0000000000001787. PMID 30239493
- [Background] Whittaker JL, Toomey CM, Woodhouse LJ, Jaremko JL, Nettel-Aguirre A, Emery CA. Association between MRI-defined osteoarthritis, pain, function and strength 3-10 years following knee joint injury in youth sport. Br J Sports Med. 2018 Jul;52(14):934-939. doi: 10.1136/bjsports-2017-097576. Epub 2017 Oct 10. PMID 29018061
- [Background] Whittaker JL, Woodhouse LJ, Nettel-Aguirre A, Emery CA. Outcomes associated with early post-traumatic osteoarthritis and other negative health consequences 3-10 years following knee joint injury in youth sport. Osteoarthritis Cartilage. 2015 Jul;23(7):1122-9. doi: 10.1016/j.joca.2015.02.021. Epub 2015 Feb 26. PMID 25725392
- [Background] Baltich J, Whittaker J, Von Tscharner V, Nettel-Aguirre A, Nigg BM, Emery C. The impact of previous knee injury on force plate and field-based measures of balance. Clin Biomech (Bristol). 2015 Oct;30(8):832-8. doi: 10.1016/j.clinbiomech.2015.06.005. Epub 2015 Jun 12. PMID 26094135
- [Background] Laudon J, Whittaker JL, Ren G, Jaremko JL, Emery CA, Krawetz RJ. Serum cartilage oligomeric matrix protein (COMP) expression in individuals who sustained a youth sport-related intra-articular knee injury 3-10 years previously and uninjured matched controls. Osteoarthritis Cartilage. 2019 Feb;27(2):286-293. doi: 10.1016/j.joca.2018.09.011. Epub 2018 Oct 11. PMID 30317002
- [Background] Ezzat AM, Whittaker JL, Toomey C, Doyle-Baker PK, Brussoni M, Emery CA. Knee confidence in youth and young adults at risk of post-traumatic osteoarthritis 3-10 years following intra-articular knee injury. J Sci Med Sport. 2018 Jul;21(7):671-675. doi: 10.1016/j.jsams.2017.11.012. Epub 2017 Nov 26. PMID 29233667
- [Background] Ezzat AM, Brussoni M, Whittaker JL, Emery CA. A qualitative investigation of the attitudes and beliefs about physical activity and post-traumatic osteoarthritis in young adults 3-10 years after an intra-articular knee injury. Phys Ther Sport. 2018 Jul;32:98-108. doi: 10.1016/j.ptsp.2018.05.001. Epub 2018 May 4. PMID 29778829
- [Background] Oiestad BE, Juhl CB, Eitzen I, Thorlund JB. Knee extensor muscle weakness is a risk factor for development of knee osteoarthritis. A systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Feb;23(2):171-7. doi: 10.1016/j.joca.2014.10.008. Epub 2014 Nov 1. PMID 25450853
- [Background] Wallace IJ, Worthington S, Felson DT, Jurmain RD, Wren KT, Maijanen H, Woods RJ, Lieberman DE. Knee osteoarthritis has doubled in prevalence since the mid-20th century. Proc Natl Acad Sci U S A. 2017 Aug 29;114(35):9332-9336. doi: 10.1073/pnas.1703856114. Epub 2017 Aug 14. PMID 28808025
- [Background] Silverwood V, Blagojevic-Bucknall M, Jinks C, Jordan JL, Protheroe J, Jordan KP. Current evidence on risk factors for knee osteoarthritis in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Apr;23(4):507-15. doi: 10.1016/j.joca.2014.11.019. Epub 2014 Nov 29. PMID 25447976
- [Background] Whittaker JL, Roos EM. A pragmatic approach to prevent post-traumatic osteoarthritis after sport or exercise-related joint injury. Best Pract Res Clin Rheumatol. 2019 Feb;33(1):158-171. doi: 10.1016/j.berh.2019.02.008. Epub 2019 Mar 14. PMID 31431269
- [Background] Feucht MJ, Cotic M, Saier T, Minzlaff P, Plath JE, Imhoff AB, Hinterwimmer S. Patient expectations of primary and revision anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2016 Jan;24(1):201-7. doi: 10.1007/s00167-014-3364-z. Epub 2014 Oct 2. PMID 25274098
- [Background] Bricca A, Wirth W, Juhl CB, Kemnitz J, Hunter DJ, Kwoh CK, Eckstein F, Culvenor AG. Moderate Physical Activity and Prevention of Cartilage Loss in People With Knee Osteoarthritis: Data From the Osteoarthritis Initiative. Arthritis Care Res (Hoboken). 2019 Feb;71(2):218-226. doi: 10.1002/acr.23791. PMID 30339323
- [Background] Janz KF, Letuchy EM, Eichenberger Gilmore JM, Burns TL, Torner JC, Willing MC, Levy SM. Early physical activity provides sustained bone health benefits later in childhood. Med Sci Sports Exerc. 2010 Jun;42(6):1072-8. doi: 10.1249/MSS.0b013e3181c619b2. PMID 19997029
- [Background] Andrade R, Pereira R, van Cingel R, Staal JB, Espregueira-Mendes J. How should clinicians rehabilitate patients after ACL reconstruction? A systematic review of clinical practice guidelines (CPGs) with a focus on quality appraisal (AGREE II). Br J Sports Med. 2020 May;54(9):512-519. doi: 10.1136/bjsports-2018-100310. Epub 2019 Jun 7. PMID 31175108
- [Background] van Melick N, van Cingel RE, Brooijmans F, Neeter C, van Tienen T, Hullegie W, Nijhuis-van der Sanden MW. Evidence-based clinical practice update: practice guidelines for anterior cruciate ligament rehabilitation based on a systematic review and multidisciplinary consensus. Br J Sports Med. 2016 Dec;50(24):1506-1515. doi: 10.1136/bjsports-2015-095898. Epub 2016 Aug 18. PMID 27539507
- [Background] Juhl C, Christensen R, Roos EM, Zhang W, Lund H. Impact of exercise type and dose on pain and disability in knee osteoarthritis: a systematic review and meta-regression analysis of randomized controlled trials. Arthritis Rheumatol. 2014 Mar;66(3):622-36. doi: 10.1002/art.38290. PMID 24574223
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Helminen HJ, Hyttinen MM, Lammi MJ, Arokoski JP, Lapvetelainen T, Jurvelin J, Kiviranta I, Tammi MI. Regular joint loading in youth assists in the establishment and strengthening of the collagen network of articular cartilage and contributes to the prevention of osteoarthrosis later in life: a hypothesis. J Bone Miner Metab. 2000;18(5):245-57. doi: 10.1007/pl00010638. No abstract available. PMID 10959613
- [Background] Logerstedt DS, Scalzitti D, Risberg MA, Engebretsen L, Webster KE, Feller J, Snyder-Mackler L, Axe MJ, McDonough CM. Knee Stability and Movement Coordination Impairments: Knee Ligament Sprain Revision 2017. J Orthop Sports Phys Ther. 2017 Nov;47(11):A1-A47. doi: 10.2519/jospt.2017.0303. PMID 29089004
- [Background] Duncan KJ, Chopp-Hurley JN, Maly MR. A systematic review to evaluate exercise for anterior cruciate ligament injuries: does this approach reduce the incidence of knee osteoarthritis? Open Access Rheumatol. 2016 Jan 8;8:1-16. doi: 10.2147/OARRR.S81673. eCollection 2016. PMID 27843365
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] O'Brien BC, Harris IB, Beckman TJ, Reed DA, Cook DA. Standards for reporting qualitative research: a synthesis of recommendations. Acad Med. 2014 Sep;89(9):1245-51. doi: 10.1097/ACM.0000000000000388. PMID 24979285
- [Background] Hemming K, Lilford R, Girling AJ. Stepped-wedge cluster randomised controlled trials: a generic framework including parallel and multiple-level designs. Stat Med. 2015 Jan 30;34(2):181-96. doi: 10.1002/sim.6325. Epub 2014 Oct 24. PMID 25346484
- [Background] Niemeijer A, Lund H, Stafne SN, Ipsen T, Goldschmidt CL, Jorgensen CT, Juhl CB. Adverse events of exercise therapy in randomised controlled trials: a systematic review and meta-analysis. Br J Sports Med. 2020 Sep;54(18):1073-1080. doi: 10.1136/bjsports-2018-100461. Epub 2019 Sep 28. PMID 31563884
- [Background] Bodkin SG, Rutherford MH, Diduch DR, Brockmeier SF, Hart JM. How Much Time Is Needed Between Serial "Return to Play" Assessments to Achieve Clinically Important Strength Gains in Patients Recovering From Anterior Cruciate Ligament Reconstruction? Am J Sports Med. 2020 Jan;48(1):70-77. doi: 10.1177/0363546519886291. Epub 2019 Nov 22. PMID 31756121
- [Background] Legare F, Stacey D, Turcotte S, Cossi MJ, Kryworuchko J, Graham ID, Lyddiatt A, Politi MC, Thomson R, Elwyn G, Donner-Banzhoff N. Interventions for improving the adoption of shared decision making by healthcare professionals. Cochrane Database Syst Rev. 2014 Sep 15;(9):CD006732. doi: 10.1002/14651858.CD006732.pub3. PMID 25222632
- [Background] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Rasmussen S. A Randomized, Controlled Trial of Total Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1597-606. doi: 10.1056/NEJMoa1505467. PMID 26488691
- [Background] Helms ER, Cronin J, Storey A, Zourdos MC. Application of the Repetitions in Reserve-Based Rating of Perceived Exertion Scale for Resistance Training. Strength Cond J. 2016 Aug;38(4):42-49. doi: 10.1519/SSC.0000000000000218. Epub 2016 Aug 3. PMID 27531969
- [Background] Truong LK, Mosewich AD, Holt CJ, Le CY, Miciak M, Whittaker JL. Psychological, social and contextual factors across recovery stages following a sport-related knee injury: a scoping review. Br J Sports Med. 2020 Oct;54(19):1149-1156. doi: 10.1136/bjsports-2019-101206. Epub 2020 Feb 14. PMID 32060141
- [Background] Li LC, Sayre EC, Xie H, Falck RS, Best JR, Liu-Ambrose T, Grewal N, Hoens AM, Noonan G, Feehan LM. Efficacy of a Community-Based Technology-Enabled Physical Activity Counseling Program for People With Knee Osteoarthritis: Proof-of-Concept Study. J Med Internet Res. 2018 Apr 30;20(4):e159. doi: 10.2196/jmir.8514. PMID 29712630
- [Background] Lewis ZH, Lyons EJ, Jarvis JM, Baillargeon J. Using an electronic activity monitor system as an intervention modality: A systematic review. BMC Public Health. 2015 Jun 24;15:585. doi: 10.1186/s12889-015-1947-3. PMID 26104189
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Tayfur B, Charuphongsa C, Morrissey D, Miller SC. Neuromuscular Function of the Knee Joint Following Knee Injuries: Does It Ever Get Back to Normal? A Systematic Review with Meta-Analyses. Sports Med. 2021 Feb;51(2):321-338. doi: 10.1007/s40279-020-01386-6. PMID 33247378
- [Background] Undheim MB, Cosgrave C, King E, Strike S, Marshall B, Falvey E, Franklyn-Miller A. Isokinetic muscle strength and readiness to return to sport following anterior cruciate ligament reconstruction: is there an association? A systematic review and a protocol recommendation. Br J Sports Med. 2015 Oct;49(20):1305-10. doi: 10.1136/bjsports-2014-093962. Epub 2015 Jun 23. PMID 26105017
- [Background] Feehan LM, Geldman J, Sayre EC, Park C, Ezzat AM, Yoo JY, Hamilton CB, Li LC. Accuracy of Fitbit Devices: Systematic Review and Narrative Syntheses of Quantitative Data. JMIR Mhealth Uhealth. 2018 Aug 9;6(8):e10527. doi: 10.2196/10527. PMID 30093371
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Bandura A. Human agency in social cognitive theory. Am Psychol. 1989 Sep;44(9):1175-84. doi: 10.1037/0003-066x.44.9.1175. PMID 2782727
- [Background] Van Der Horst K, Paw MJ, Twisk JW, Van Mechelen W. A brief review on correlates of physical activity and sedentariness in youth. Med Sci Sports Exerc. 2007 Aug;39(8):1241-50. doi: 10.1249/mss.0b013e318059bf35. PMID 17762356
- [Background] Thomee P, Wahrborg P, Borjesson M, Thomee R, Eriksson BI, Karlsson J. Self-efficacy, symptoms and physical activity in patients with an anterior cruciate ligament injury: a prospective study. Scand J Med Sci Sports. 2007 Jun;17(3):238-45. doi: 10.1111/j.1600-0838.2006.00557.x. Epub 2006 Jun 15. PMID 16774652
- [Background] Collins NJ, Prinsen CA, Christensen R, Bartels EM, Terwee CB, Roos EM. Knee Injury and Osteoarthritis Outcome Score (KOOS): systematic review and meta-analysis of measurement properties. Osteoarthritis Cartilage. 2016 Aug;24(8):1317-29. doi: 10.1016/j.joca.2016.03.010. Epub 2016 Mar 21. PMID 27012756
- [Background] Chatman AB, Hyams SP, Neel JM, Binkley JM, Stratford PW, Schomberg A, Stabler M. The Patient-Specific Functional Scale: measurement properties in patients with knee dysfunction. Phys Ther. 1997 Aug;77(8):820-9. doi: 10.1093/ptj/77.8.820. PMID 9256870
- [Background] Amireault S, Godin G. The Godin-Shephard leisure-time physical activity questionnaire: validity evidence supporting its use for classifying healthy adults into active and insufficiently active categories. Percept Mot Skills. 2015 Apr;120(2):604-22. doi: 10.2466/03.27.PMS.120v19x7. Epub 2015 Mar 23. PMID 25799030
- [Background] Smith D, Harvey P, Lawn S, Harris M, Battersby M. Measuring chronic condition self-management in an Australian community: factor structure of the revised Partners in Health (PIH) scale. Qual Life Res. 2017 Jan;26(1):149-159. doi: 10.1007/s11136-016-1368-5. Epub 2016 Jul 18. PMID 27432251
- [Background] Kvist J, Ek A, Sporrstedt K, Good L. Fear of re-injury: a hindrance for returning to sports after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2005 Jul;13(5):393-7. doi: 10.1007/s00167-004-0591-8. Epub 2005 Feb 10. PMID 15703963
- [Background] Mitchell I, Evans L, Rees T, Hardy L. Stressors, social support, and tests of the buffering hypothesis: effects on psychological responses of injured athletes. Br J Health Psychol. 2014 Sep;19(3):486-508. doi: 10.1111/bjhp.12046. Epub 2013 Apr 27. PMID 23621677
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326
- [Background] Canty-Mitchell J, Zimet GD. Psychometric properties of the Multidimensional Scale of Perceived Social Support in urban adolescents. Am J Community Psychol. 2000 Jun;28(3):391-400. doi: 10.1023/A:1005109522457. PMID 10945123
- [Background] Freeman P, Coffee P, Rees T. The PASS-Q: the perceived available support in sport questionnaire. J Sport Exerc Psychol. 2011 Feb;33(1):54-74. doi: 10.1123/jsep.33.1.54. PMID 21451171
- [Background] Fischer F, Fink C, Herbst E, Hoser C, Hepperger C, Blank C, Gfoller P. Higher hamstring-to-quadriceps isokinetic strength ratio during the first post-operative months in patients with quadriceps tendon compared to hamstring tendon graft following ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2018 Feb;26(2):418-425. doi: 10.1007/s00167-017-4522-x. Epub 2017 Mar 21. PMID 28324151
- [Background] Abourezk MN, Ithurburn MP, McNally MP, Thoma LM, Briggs MS, Hewett TE, Spindler KP, Kaeding CC, Schmitt LC. Hamstring Strength Asymmetry at 3 Years After Anterior Cruciate Ligament Reconstruction Alters Knee Mechanics During Gait and Jogging. Am J Sports Med. 2017 Jan;45(1):97-105. doi: 10.1177/0363546516664705. Epub 2016 Oct 1. PMID 27590173
- [Background] Kline PW, Jacobs CA, Duncan ST, Noehren B. Rate of torque development is the primary contributor to quadriceps avoidance gait following total knee arthroplasty. Gait Posture. 2019 Feb;68:397-402. doi: 10.1016/j.gaitpost.2018.12.019. Epub 2018 Dec 16. PMID 30594013
- [Background] Reid KF, Price LL, Harvey WF, Driban JB, Hau C, Fielding RA, Wang C. Muscle Power Is an Independent Determinant of Pain and Quality of Life in Knee Osteoarthritis. Arthritis Rheumatol. 2015 Dec;67(12):3166-73. doi: 10.1002/art.39336. PMID 26315282
- [Background] Kline PW, Morgan KD, Johnson DL, Ireland ML, Noehren B. Impaired Quadriceps Rate of Torque Development and Knee Mechanics After Anterior Cruciate Ligament Reconstruction With Patellar Tendon Autograft. Am J Sports Med. 2015 Oct;43(10):2553-8. doi: 10.1177/0363546515595834. Epub 2015 Aug 14. PMID 26276828
- [Background] Cobian DG, Koch CM, Amendola A, Williams GN. Knee Extensor Rate of Torque Development Before and After Arthroscopic Partial Meniscectomy, With Analysis of Neuromuscular Mechanisms. J Orthop Sports Phys Ther. 2017 Dec;47(12):945-956. doi: 10.2519/jospt.2017.7310. Epub 2017 Oct 9. PMID 28992769
- [Background] Davis HC, Troy Blackburn J, Ryan ED, Luc-Harkey BA, Harkey MS, Padua DA, Pietrosimone B. Quadriceps rate of torque development and disability in individuals with anterior cruciate ligament reconstruction. Clin Biomech (Bristol). 2017 Jul;46:52-56. doi: 10.1016/j.clinbiomech.2017.04.011. Epub 2017 Apr 28. PMID 28511105
- [Background] Hunt MA, Charlton JM, Esculier JF. Osteoarthritis year in review 2019: mechanics. Osteoarthritis Cartilage. 2020 Mar;28(3):267-274. doi: 10.1016/j.joca.2019.12.003. Epub 2019 Dec 23. PMID 31877382
- [Background] Wellsandt E, Axe MJ, Snyder-Mackler L. Poor Performance on Single-Legged Hop Tests Associated With Development of Posttraumatic Knee Osteoarthritis After Anterior Cruciate Ligament Injury. Orthop J Sports Med. 2018 Nov 26;6(11):2325967118810775. doi: 10.1177/2325967118810775. eCollection 2018 Nov. PMID 30505875
- [Background] Losciale JM, Bullock G, Cromwell C, Ledbetter L, Pietrosimone L, Sell TC. Hop Testing Lacks Strong Association With Key Outcome Variables After Primary Anterior Cruciate Ligament Reconstruction: A Systematic Review. Am J Sports Med. 2020 Feb;48(2):511-522. doi: 10.1177/0363546519838794. Epub 2019 May 7. PMID 31063403
- [Background] Davies WT, Myer GD, Read PJ. Is It Time We Better Understood the Tests We are Using for Return to Sport Decision Making Following ACL Reconstruction? A Critical Review of the Hop Tests. Sports Med. 2020 Mar;50(3):485-495. doi: 10.1007/s40279-019-01221-7. PMID 31745732
- [Background] Reid A, Birmingham TB, Stratford PW, Alcock GK, Giffin JR. Hop testing provides a reliable and valid outcome measure during rehabilitation after anterior cruciate ligament reconstruction. Phys Ther. 2007 Mar;87(3):337-49. doi: 10.2522/ptj.20060143. Epub 2007 Feb 20. PMID 17311886
- [Background] Talma H, Chinapaw MJ, Bakker B, HiraSing RA, Terwee CB, Altenburg TM. Bioelectrical impedance analysis to estimate body composition in children and adolescents: a systematic review and evidence appraisal of validity, responsiveness, reliability and measurement error. Obes Rev. 2013 Nov;14(11):895-905. doi: 10.1111/obr.12061. Epub 2013 Jul 12. PMID 23848977
- [Background] Leahy S, O'Neill C, Sohun R, Jakeman P. A comparison of dual energy X-ray absorptiometry and bioelectrical impedance analysis to measure total and segmental body composition in healthy young adults. Eur J Appl Physiol. 2012 Feb;112(2):589-95. doi: 10.1007/s00421-011-2010-4. Epub 2011 May 26. PMID 21614505
- [Background] Coyne IT. Sampling in qualitative research. Purposeful and theoretical sampling; merging or clear boundaries? J Adv Nurs. 1997 Sep;26(3):623-30. doi: 10.1046/j.1365-2648.1997.t01-25-00999.x. PMID 9378886
- [Background] Schoenfeld D. Statistical considerations for pilot studies. Int J Radiat Oncol Biol Phys. 1980 Mar;6(3):371-4. doi: 10.1016/0360-3016(80)90153-4. No abstract available. PMID 7390914
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Wilson PM, Petticrew M, Calnan MW, Nazareth I. Disseminating research findings: what should researchers do? A systematic scoping review of conceptual frameworks. Implement Sci. 2010 Nov 22;5:91. doi: 10.1186/1748-5908-5-91. PMID 21092164
- [Derived] Whittaker JL, Truong LK, Losciale JM, Silvester-Lee T, Miciak M, Pajkic A, Le CY, Hoens AM, Mosewich A, Hunt MA, Li LC, Roos EM. Efficacy of the SOAR knee health program: protocol for a two-arm stepped-wedge randomized delayed-controlled trial. BMC Musculoskelet Disord. 2022 Jan 25;23(1):85. doi: 10.1186/s12891-022-05019-z. PMID 35078446